CLINICAL TRIAL: NCT06109298
Title: The Effect of Cold Spray and Ice Applied During Intravenous Access on Pain and Fear in Children Aged 7-15 Years in Pediatric Emergency Unit
Brief Title: The Effect of Cold Spray and Ice Applied During Intravenous Access on Pain and Fear i in Pediatric Emergency Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Duygu Sonmez Duzkaya, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 347
Record Dates: First submitted 2023-10-24; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Children, Only; Pain; Emergencies
Keywords: ıce pack; cold spray; fear; pain
MeSH Terms: conditions — Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First study group (Experimental): Before performing intravenous intervention, cold spray was applied for 5 seconds at a distance of 15 cm to an area of approximately 5 cm2 at the site of the procedure. After tourniquet fixation and subsequent skin disinfection for 60 seconds, the nurse researcher performed intravenous administration.
  Interventions: Other: Cold spray
- Second study group (Experimental): Before the intravenous intervention, refrigerated gel ice was applied for 5 minutes at 2 cm above the area to be treated. After that, the nurse removed the gel ice from the procedure area, a tourniquet was applied, and skin disinfection was performed for 60 seconds. The nurse researcher performed intravenous administration.
  Interventions: Other: Refrigerated gel ice
- Control group (No Intervention): No pharmacologic or nonpharmacologic application was performed. The researcher performed intravenous access after skin disinfection by the nurse.

INTERVENTIONS:
Other: Cold spray — Cold spray was applied for 5 seconds at a distance of 15 cm to an area of approximately 5 cm2 at the site of the procedu
  Arms: First study group
Other: Refrigerated gel ice — Refrigerated gel ice was applied for 5 minutes at 2 cm above the area to be treated.
  Arms: Second study group

SUMMARY:
Many strategies have been developed for the prevention of to prevent procedural pain in pediatric emergency units where nurses play a vital role in patient comfort.Easy-to-use and inexpensive nonpharmacologic analgesic methods are important in emergency units.This study was conducted to determine the effect of cold spray and ice applied during venipuncture on the level of fear and pain in children ages 7-15. This randomized, controlled experimental study was conducted in the Pediatric Emergency Clinic of Istanbul Gaziosmanpaşa Training and Research Hospital between November 2021 7 and April 2022. The study was conducted with 96 children between the ages of 7 and 15 (cold spray group, ice group, and control group) who were scheduled to have venous access in the pediatric emergency clinic and met the sampling criteria.

The Pediatric Emergency Clinic consists of 10 beds. Patients with complaints such as fever, vomiting, diarrhea, and seizures comprise the majority of those admitted to the clinic. In the Pediatric Emergency Clinic, intravenous interventions were performed in the injection room.

DETAILED DESCRIPTION:
This study aimed to determine the effect of cold spray and ice applied during venipuncture procedures on pain and fear in 67 children ages 7-15 admitted to the pediatric emergency unit.

Materials and Methods Setting This randomized, controlled experimental study was conducted in the Pediatric Emergency Clinic of Istanbul Gaziosmanpaşa Training and Research Hospital between November 2021 7 and April 2022. The Pediatric Emergency Clinic consists of 10 beds. Patients with complaints such as fever, vomiting, diarrhea, and seizures comprise the majority of those admitted to the clinic. In the Pediatric Emergency Clinic, intravenous interventions were performed in the injection room.

Sample The study's population comprised children ages 7-15 treated in the Pediatric Emergency Department of Gaziosmanpaşa Training and Research Hospital. The sample consisted of children undergoing intravenous access in line with the inclusion criteria. According to the power analysis for the sample size in line with the literatüre the power of the sample was calculated with the G*Power 3.1 program. With a Type I error of 0.05 and a test power of 0.80 (α= 0.05, 1-β= 0.80), the minimum sample size was calculated as children (30 children in 83 each group). The study was completed with 96 children, including 32 children in the study and control groups, taking into account the losses that might occur from the sample for any reason during the study period.

Allocation In the study, 96 children in the sample will randomly assigned to the control (n=32), ice (n=32), and spray groups (n=32). Random assignment will ensured by using a computer program to determine the group of children (https://www.randomlists.com/team-generator).

Data Collection Before starting the study, the families of the children were informed of the purpose, plan, duration, and how the data would be used. Written consent was obtained in light of the principle of willingness and voluntariness through the Voluntary Information and Consent Form. Pediatric patients included in the study were divided into three groups: cold spray, ice, and control. Environmental conditions were organized the same way in all three groups, and at least one parent was ensured to stay with each child. The study was conducted with a nurse performing intravenous intervention and a nurse researcher.

IV Catheter placement IV placement was performed using 24-gauge catheters appropriate in size for the age of the children and took an average of 3 minutes. The observer nurse evaluated the children in all groups before and after the procedure by filling out the data collection form and measuring the child's pain and fear assessment scales. The pain and fear scales were also evaluated by the child and parent. In all groups, IV insertion was performed by the same nurse following the procedure steps.

* First study group: Before performing intravenous intervention, cold spray was applied for 5 seconds at a distance of 15 cm to an area of approximately 5 cm2 at the site of the procedure. After tourniquet fixation and subsequent skin disinfection for 60 seconds, the nurse researcher performed intravenous administration.
* Second study group: Before the intravenous intervention, refrigerated gel ice was applied for 5 minutes at 2 cm above the area to be treated. After that, the nurse removed the gel ice from the procedure area, a tourniquet was applied, and skin disinfection was performed for 60 seconds. The nurse researcher performed intravenous administration.
* Control group: No pharmacologic or nonpharmacologic application was performed. The researcher performed intravenous access after skin disinfection by the nurse.

ETHICAL CONSIDERATION Written permission were obtained from the ethics committee of Gaizosmanpaşa Training and Research Hospital to collect the data before the study (No: 347, Date: 20.10.2021). The rules of the Declaration of Helsinki were followed throughout the study. Verbal and written informed consent was obtained from the families of pediatric patients who agreed to participate in the study. After patients entered the pediatric emergency clinic in accordance with the sample selection criteria, the parents were explained the purpose of the research, that their personal information would remain confidential, and that their privacy would be respected.

STATISTICAL ANALYSIS Statistical analyses were performed using R vers. 2.15.3 program Minimum, maximum, mean, standard deviation, median, first quartile, third quartile, frequency, and percentage were used to report the study data. The Shapiro-Wilk test and graphical analysis were used to evaluate the compliance of quantitative data with normal distribution. A dependent groups t-test was used to compare the values before and after the intervention. An independent groups t-test was used to evaluate normally distributed variables between two groups. One-way analysis of variance was used in the evaluations of variables with normal distribution between more than two groups. The Mann-Whitney U test evaluated variables that did not show normal distribution between the two groups. The Kruskal-Wallis test was used in the evaluations of variables that did not show normal distribution between more than two groups. Pearson correlation analysis was used to determine the relationship between quantitative variables. The Pearson chi-square test, Fisher-Freeman-Halton exact test, and Fisher's exact test were used to compare qualitative variables. Statistical significance was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the study were 7-15 years old
* volunteered to participate
* Had no chronic diseases, mental or neurological disabilities, neurodevelopmental impairments, or life threatening conditions (sepsis, shock, respiratory/cardiogenic arrest, etc.).

Exclusion Criteria:

* Children who had taken any analgesic medication before presentation to the emergency department
* had undergone multiple attempts for vascular access

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Data Collection Form | 1 day
  The data collection form was prepared by reviewing the literature on the subject. It consisted of a total of 15 questions, including questions about the child's and family's descriptive characteristics (such as age and gender), the reason for going to the emergency room, and complaints, such as previous emergency room visits
Child Fear Scale | 1 day
  The Child Fear Scale is used to assess the anxiety levels of children with five face shapes scored between 0-4: 0 = no anxiety, and 4 = severe anxiety. The scale can be evaluated by both the child and the researcher before, during, and after the intervention.
Visual Analog Scale | 1 day
  The VAS is the most frequently used scale in pain studies. In children over 7 years of age, it is frequently used because it is common and easy. The VAS is a pain scale with numbers from 1 to 10, equally spaced on a 10 cm horizontal ruler. Children being assessed are asked to choose a pain value between 1 and 10 on this ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- [Background] Su HC, Hsieh CW, Lai NM, Chou PY, Lin PH, Chen KH. Using Vibrating and Cold Device for Pain Relieves in Children: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Pediatr Nurs. 2021 Nov-Dec;61:23-33. doi: 10.1016/j.pedn.2021.02.027. Epub 2021 Mar 16. PMID 33735633
- [Background] Bergomi P, Scudeller L, Pintaldi S, Dal Molin A. Efficacy of Non-pharmacological Methods of Pain Management in Children Undergoing Venipuncture in a Pediatric Outpatient Clinic: A Randomized Controlled Trial of Audiovisual Distraction and External Cold and Vibration. J Pediatr Nurs. 2018 Sep-Oct;42:e66-e72. doi: 10.1016/j.pedn.2018.04.011. Epub 2018 May 1. PMID 29728296
- [Background] Canbulat Sahiner N, Inal S, Sevim Akbay A. The effect of combined stimulation of external cold and vibration during immunization on pain and anxiety levels in children. J Perianesth Nurs. 2015 Jun;30(3):228-35. doi: 10.1016/j.jopan.2014.05.011. PMID 26003770
- [Background] Inal S, Kelleci M. The Effect of External Thermomechanical Stimulation and Distraction on Reducing Pain Experienced by Children During Blood Drawing. Pediatr Emerg Care. 2020 Feb;36(2):66-69. doi: 10.1097/PEC.0000000000001264. PMID 28885392
- [Background] Potts DA, Davis KF, Elci OU, Fein JA. A Vibrating Cold Device to Reduce Pain in the Pediatric Emergency Department: A Randomized Clinical Trial. Pediatr Emerg Care. 2019 Jun;35(6):419-425. doi: 10.1097/PEC.0000000000001041. PMID 28121978
- [Background] Redfern RE, Micham J, Sievert D, Chen JT. Effects of Thermomechanical Stimulation During Intravenous Catheter Insertion in Adults: A Prospective Randomized Study. J Infus Nurs. 2018 Sep/Oct;41(5):294-300. doi: 10.1097/NAN.0000000000000294. PMID 30188451
- [Background] Zhu Y, Peng X, Wang S, Chen W, Liu C, Guo B, Zhao L, Gao Y, Wang K, Lou F. Vapocoolant spray versus placebo spray/no treatment for reducing pain from intravenous cannulation: A meta-analysis of randomized controlled trials. Am J Emerg Med. 2018 Nov;36(11):2085-2092. doi: 10.1016/j.ajem.2018.03.068. Epub 2018 Mar 27. PMID 30253890
- [Background] Mu Y, Wang L. Standardized post-catheter nursing intervention reduces incidence of catheter complications in the disabled elderly and improves their quality of life. Am J Transl Res. 2021 Nov 15;13(11):12957-12964. eCollection 2021. PMID 34956511